CLINICAL TRIAL: NCT04340297
Title: Randomized Double-Blind Clinical Trial of Tongjiang Theory and Syndrome Differentiation Serial Prescriptions Combined With Proton Pump Inhibitors(PPIs)Descending Ladder Withdrawal for the Treatment of Nonerosive Reflux Disease.
Brief Title: Tongjiang Series Prescription Combined With PPIs Descending Ladder Withdrawal in Treating Nonerosive Reflux Disease
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xiyuan Hospital of China Academy of Chinese Medical Sciences (Other)
Collaborators: Guangdong Provincial Hospital of Traditional Chinese Medicine (Other); Wuhan No.1 Hospital (Other); The First Affiliated Hospital of Tianjin University of Traditional Chinese Medicine (Other); Traditional Chinese Medicine Hospital of KUNSHAN (Unknown); Liuzhou Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019YFC1709604
Record Dates: First submitted 2020-04-01; First posted 2020-04-09 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Nonerosive Reflux Disease
Keywords: Traditional Chinese medicine; Tongjiang series prescription; Randomized controlled trial

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Tongjiang granules are taken orally in liver-stomach depression-heat syndrome, Jianpi Qinghua granules are taken orally in spleen deficiency damp-heat syndrome, Wenpi Qingwei granules are taken orally in cold-heat complicated syndrome, one bag per time, 3 times a day and 1 hour after a meal. At the same time, it was combined with acid inhibitors to reduce the steps of withdrawal treatment: in the 1-2 weeks, acid inhibitor (PPI) was reduced from the dose before entering the group to half of the dose, once a day, before going to bed; in the 3-4 weeks, acid inhibitor was changed from PPI to famotidine tablets, 20mg each time, before going to bed; in the 5-6 weeks, all acid inhibitors were stopped.
  Interventions: Drug: Tongjiang series prescription(Tongjiang granules, Jianpi Qinghua granules and Wenpi Qingwei granules); Drug: Acid inhibitors
- Control group (Placebo Comparator): Tongjiang placebo granules are taken orally by patients with liver-stomach depression-heat syndrome, Jianpi Qinghua placebo granules are taken orally by patients with spleen deficiency damp-heat syndrome, Wenpi Qingwei placebo granules are taken orally by patients with cold-heat complicated syndrome, 1 bag per time, 3 times a day and 1 hour after a meal. At the same time, it was combined with acid inhibitors to reduce the steps of withdrawal treatment: in the 1-2 weeks, acid inhibitor (PPI) was reduced from the dose before entering the group to half of the dose, once a day, before going to bed; in the 3-4 weeks, acid inhibitor was changed from PPI to famotidine tablets, 20mg each time, before going to bed; in the 5-6 weeks, all acid inhibitors were stopped.
  Interventions: Drug: Acid inhibitors; Drug: Placebo

INTERVENTIONS:
Drug: Tongjiang series prescription(Tongjiang granules, Jianpi Qinghua granules and Wenpi Qingwei granules) — According to the syndrome differentiation of TCM, Tongjiang granules are taken orally by patients with liver-stomach depression-heat syndrome, Jianpi Qinghua granules are taken orally by patients with spleen deficiency damp-heat syndrome, Wenpi Qingwei granules are taken orally by patients with cold-heat complicated syndrome, 1 bag per time, 3 times a day and 1 hour after a meal.
  Arms: Experimental group
Drug: Acid inhibitors — In the 1-2 weeks, acid inhibitor (PPI) was reduced from the dose before entering the group to half of the dose, once a day, before going to bed; in the 3-4 weeks, acid inhibitor was changed from PPI to famotidine tablets, 20mg each time, before going to bed; in the 5-6 weeks, all acid inhibitors were stopped.
Drug: Placebo — Tongjiang granules placebo , Jianpi Qinghua granules placebo and Wenpi Qingwei granules placebo. The above three kinds of granulated placebo are respectively made of the simulation containing the low dose original prescription. Taking method is the same as Tongjiang series prescription.
  Arms: Control group

SUMMARY:
Nonerosive Reflux Disease (NERD) is a common refractory gastrointestinal disease. Proton Pump Inhibitors (PPIs), the preferred drug, have poor response, single target and poor acid inhibition effect in some patients in clinical application. Long-term use of PPI can lead to many side effects, even dependency. The main Traditional Chinese Medicine (TCM)syndrome types of NERD are liver-stomach depression-heat syndrome, spleen deficiency damp-heat syndrome and cold-heat complicated syndrome. TCM syndrome differentiation treatment has the advantages of overall regulation and individualized treatment. The purpose of this study is to evaluate the safety and efficacy advantages of syndrome differentiation series prescription combined with PPIs descending ladder withdrawal in the treatment of patients who use PPIs for a long time that can not stop, and to solve the problems of multiple side effects and dependency caused by long-term use of PPIs.

DETAILED DESCRIPTION:
Nonerosive Reflux Disease (NERD) accounts for about 70% of Gastroesophageal Reflux Disease (GERD), which is a common refractory gastrointestinal disease. Proton Pump Inhibitors (PPIs), the preferred treatment, have the following problems in clinical use: about 50% of patients respond to PPIs only partially or not at all; PPIs has a single target, and the effect of acid suppression alone is poor; long term use of PPIs can lead to dyspepsia, fundic gland polyp, atrophic gastritis, intestinal flora disorders, and even dependency. Liver-stomach depression-heat syndrome, spleen deficiency damp-heat syndrome and cold-heat complicated syndrome account for 80%-91% of NERD's Traditional Chinese Medicine (TCM) syndrome. TCM syndrome differentiation treatment has the advantages of overall regulation and individualized treatment, but it lacks high-level evidence-based medicine evidence. On the basis of previous work, the project plans to establish sub centers in 6 Chinese hospitals, including 180 patients with NERD who meet the requirements to carry out a multicenter, randomized, double-blind, placebo-controlled clinical study, in which 90 subjects in the experimental group received the treatment of syndrome differentiation series of prescriptions combined with PPIs descending ladder withdrawal, and 90 subjects in the control group received the treatment of placebo combined with PPIs descending ladder withdrawal. The therapeutic effects were evaluated from the following aspects: the VAS score of reflow and heartburn, the rate of discontinuation of antacids, the rate of recurrence of NERD symptoms, the score of TCM syndromes and the improvement of gastrointestinal function. The purpose of this study is to evaluate the efficacy advantage and safety of Tongjiang series prescription combined with PPIs descending ladder withdrawal compared with PPIs descending ladder withdrawal alone for patients who use PPIs for a long time that can not stop, so as to obtain evidence-based medical evidence of high-quality TCM syndrome differentiation treatment of NERD, and form an effective and popularized treatment plan to solve the problems of various side effects and dependency caused by long-term use of PPIs.

ELIGIBILITY:
Inclusion Criteria:

* 1. It meets the diagnostic criteria of nonerosive reflex disease(NERD)
* 2. Patients with PPIs who are effective for more than 8 weeks and relapse after discontinuation
* 3. Age between 18 and 70 years old
* 4. It meets the diagnostic criteria of liver-stomach depression-heat syndrome, spleen deficiency damp-heat syndrome and cold-heat complicated syndrome of traditional Chinese medicine
* 5. Patients have informed consent and are willing to receive corresponding treatment

Exclusion Criteria:

* 1. Patients with active peptic ulcer, gastrointestinal hemorrhage, severe dysplasia of gastric mucosa or suspected malignant change, achalasia or postoperative achalasia
* 2. There are other organic diseases of the digestive system (such as acute and chronic pancreatitis, cirrhosis, etc.), or systemic diseases that affect the gastrointestinal motility, such as hyperthyroidism, diabetes mellitus over 10 years, chronic renal insufficiency, spirit (the score of SAS and SDS shows severe anxiety or depression), nervous system diseases, etc
* 3. Patients with severe organ diseases such as heart, liver and kidney (such as ALT, AST more than 2 times of normal value), hematopoietic system diseases and tumors
* 4. Pregnant and lactating women
* 5. Patients with history of nervous system disease and mental disease
* 6. People with a history of allergies to all the test drugs
* 7. Subjects who are participating in other clinical trials or have participated in other clinical trials within 4 weeks

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2020-06-15 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes of visual analogue (VAS) scores of reflow, heartburn and other major symptoms | 6 weeks during treatment period, 4 weeks during follow-up period
  During the period of taking medicine, the patients recorded the reflow and heartburn attacks (attack times and duration) within 24 hours every day on the symptom diary card, and VAS scores were performed on the reflow and heartburn symptoms. The average score of each symptom in the past week was calculated. The decrease rate of symptom score ≥ 50% after weekly treatment was recorded as response, and the number of response weeks was more than 50% of the whole treatment period, which was considered effective.
Discontinuation rate of acid inhibitors | 6 weeks of treatment
  Discontinuation rate of acid inhibitors = Number of drug discontinuation/ Total number of people in each group
The change of recurrence rate of main symptoms in Nonerosive Reflux Disease | 6 weeks of treatment, 4 weeks during follow-up period
  The recurrence rate of the main symptoms, such as heartburn and reflux, was evaluated respectively. The recurrence rate = Number of symptom recurrence / Number of drug discontinuation.

SECONDARY OUTCOMES:
Changes in secondary symptom scores | 6 weeks during treatment period, 4 weeks during follow-up period
  Secondary symptoms such as non cardiogenic chest pain, epigastric pain, burning sensation of epigastrium, belching, cough, asthma and foreign body sensation in pharynx were recorded and scored. Symptom frequency: none: 0 point; < 1 day / week: 1 point; 1 day / week: 2 points; 2-3 days / week: 3 points; 4-5 days / week: 4 points; 6-7 days / week: 5 points. Symptom degree: the symptom is not obvious, requiring the doctor's warning: 1 point; the symptom is obvious, affecting daily life, occasionally taking medicine: 3 points; the symptom is very obvious, affecting daily life, requiring long-term taking medicine: 5 points; between 1 point and 3 points, 2 points; between 3 points and 5 points, 4 points.
Changes of Traditional Chinese Medicine syndrome score | Baseline, 2 weeks, 4 weeks and 6 weeks during treatment period, 2 weeks and 4 weeks during follow-up period
  Before and after treatment and during follow-up, TCM syndrome scores were recorded. Symptoms are divided into four grades: asymptomatic; mild: mild, not affecting daily life; moderate: moderate, partially affecting daily life; severe: severe, affecting daily life, hard to stick to work. According to the weight of syndrome main and secondary symptoms, the main symptoms are 0 points, 2 points, 4 points and 6 points respectively, and the secondary symptoms are 0 points, 1 point, 2 points and 3 points respectively.
Changes of Gastroesophageal Reflux Disease-Health Related Quality of Life (GERD-HRQL) scale scores | Baseline, 2 weeks, 4 weeks and 6 weeks during treatment period, 2 weeks and 4 weeks during follow-up period
  The gastroesophageal Reflux Disease-Health Related Quality of Life (GERD-HRQL) scale score was evaluated before and after treatment and during follow-up. The scoring standard is the same as the international standard.
The change of the score of chronic gastrointestinal disease patient reported outcome (PRO) scale | Baseline, 2 weeks, 4 weeks and 6 weeks during treatment period, 2 weeks and 4 weeks during follow-up period
  Before and after treatment and during the follow-up period, the chronic gastrointestinal disease patient reported outcome (PRO) scale score was evaluated. The scoring standard is the same as the international standard.
The change of Self-rating anxiety scale (SAS) score | Baseline, 2 weeks, 4 weeks and 6 weeks during treatment period, 2 weeks and 4 weeks during follow-up period
  The anxiety was evaluated before and after treatment and during follow-up. The scoring standard is the same as the international standard.
The change of Self-rating depression scale (SDS) score | Baseline, 2 weeks, 4 weeks and 6 weeks during treatment period, 2 weeks and 4 weeks during follow-up period
  The depression was evaluated before and after treatment and during follow-up. The scoring standard is the same as the international standard.

CONTACTS AND LOCATIONS:
Overall Officials: Xudong Tang, M.D., Principal Investigator — China Academy of Chinese Medical Sciences
Locations (1):
- Xiyuan Hospital of China Academy of Chinese Medical Sciences, Beijing, China

REFERENCES:
- [Derived] Li X, Wu H, Zhang B, Chen T, Shi X, Ma J, Zhang J, Tang X, Wang F. Traditional Chinese medicine based on Tongjiang methodology combined with proton pump inhibitor (PPI) step-down in treating non-erosive reflux disease: a study protocol for a multicentered, randomized controlled clinical trial. Trials. 2022 Oct 18;23(1):879. doi: 10.1186/s13063-022-06811-x. PMID 36258217